CLINICAL TRIAL: NCT05470049
Title: A Phase II, Randomized, Double-Blind Study of the Combination of SHR8554 Injection and SHR0410 Injection for the Treatment of Pain After Abdominal Surgery.
Brief Title: A Clinical Study of the Combination of SHR8554 Injection and SHR0410 Injection for the Treatment of Pain After Abdominal Surgery.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR8554/SHR0410-201
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A: SHR8554 Injection and SHR0410 Injection (Experimental)
  Interventions: Drug: SHR8554 Injection and SHR0410 Injection
- Treatment group B: SHR8554 Injection and SHR0410 Injection (Experimental)
  Interventions: Drug: SHR8554 Injection and SHR0410 Injection
- Treatment group C: SHR8554 Injection and Placebo for SHR0410 Injection (Placebo Comparator)
  Interventions: Drug: SHR8554 Injection and Placebo for SHR0410 Injection

INTERVENTIONS:
Drug: SHR8554 Injection and SHR0410 Injection — Treatment group A: SHR8554 Injection and SHR0410 Injection; high dose
  Arms: Treatment group A: SHR8554 Injection and SHR0410 Injection
Drug: SHR8554 Injection and SHR0410 Injection — Treatment group B: SHR8554 Injection and SHR0410 Injection; low dose
  Arms: Treatment group B: SHR8554 Injection and SHR0410 Injection
Drug: SHR8554 Injection and Placebo for SHR0410 Injection — Treatment group C: SHR8554 Injection and Placebo for SHR0410 Injection
  Arms: Treatment group C: SHR8554 Injection and Placebo for SHR0410 Injection

SUMMARY:
The primary objective is to evaluate the analgesic efficacy of the combination of SHR8554 injection and SHR0410 injection compared with SHR8554 injection in patients with acute postoperative pain following abdominal surgery

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Subjects requiring elective general anesthesia abdominal surgery
3. Conform to the ASA Physical Status Classification

Exclusion Criteria:

1. Subjects with a history of difficult airway
2. Subjects with a history of reflux esophagitis
3. Subjects with a history of mental illness
4. Subjects with poor blood pressure control
5. Random blood glucose ≥11.1mmol/L
6. Subjects with abnormal liver function
7. allergies to opioids and other medications that may be used during the trial
8. The investigators determined that other conditions were inappropriate for participation in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
the Sum of Pain Intensity Differences in Pain Score Over 24 Hours | 24-hours
  Pain intensity will be evaluated using an 11-point (0-10) Numeric Pain Rating Scale (NPRS), with higher numbers indicating a higher pain intensity, administered over 24 hours. Time weighted average change from baseline is calculated using the following: time weighted sum of pain intensity differences (SPID) divided by a constant (24 hours) to yield values on the 0-10 NPRS.

SECONDARY OUTCOMES:
the Sum of Pain Intensity Differences in Pain Score Over 6、12、12-24 Hours | 6-hours、12-hours、12-24 hours
  time weighted sum of pain intensity differences (SPID) divided by a constant (6、12、12-24 hours) to yield values on the 0-10 NPRS.
Time of first use of remedial analgesic medication | 24-hours
  The first time to use remedial analgesic medication for injection
Cumulative use of remedial analgesics from 0h to 24h | 24-hours
  Cumulative use of remedial analgesic medication
Participant ' satisfaction score for analgesia treatment | 24-hours
  Participants recalled the postoperative analgesia effect and rated their satisfaction on a scale of 0 to 10, with 0 representing dissatisfied and 10 representing very satisfied.
Investigator satisfaction score for analgesia treatment | 24-hours
  Postoperative analgesia was evaluated by investigators.The scale ranges from 0 to 10, with 0 being dissatisfied and 10 being very satisfied.

IPD SHARING:
Plan to Share IPD: Undecided